CLINICAL TRIAL: NCT03766711
Title: FEATHERS 2.0: Functional Engagement in Assistive Therapy Through Exercise Robotics v2.0
Brief Title: VR Error Augmentation for Bimanual Task Exercise
Acronym: FEATHERSv2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Kids Brain Health Network (Unknown)
Responsible Party: Principal Investigator, Hendrik F. Machiel Van der Loos, Associate Professor, Dept. Mechanical Engineering, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H17-01126
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Hemiparesis; Cerebral Palsy; Acquired Brain Injury
Keywords: Bimanual Task; Motor Adaptation
MeSH Terms: conditions — Paresis; Cerebral Palsy; Brain Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant intervention arm will be randomized and they will not be told which whether the treatment is being applied in the current set. However, they will be instructed of the task goal at the beginning of the session and will be told that we will be modifying visual feedback to help improve reaching symmetry in some manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual - Augmented (Experimental): Reaching task as a physical therapy intervention. First with 1:1 visual feedback, then with augmented forward symmetry.
  Interventions: Other: Physical Therapy
- Augmented - Actual (Experimental): Reaching task as a physical therapy intervention. First with augmented forward symmetry, then with 1:1 visual feedback.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Repetitive bimanual task training for upper limb motor function recovery.

SUMMARY:
This project is a continuing study from the FEATHERS project (NCT02290353) which focuses on developing novel home therapy program for persons with hemiparesis. This study will focus on examining motor behaviour and adaptation in neurodevelopmental hemiparesis (cerebral palsy, acquired brain injury (ABI)). New algorithms for motion control involved in encouraging active movement are developed and will be tested, but the study has the same therapeutic goal and focus as the original FEATHERS project of creating an engaging at-home bimanual upper limb training program. By incorporating existing gaming technology, we hope to discover novel ways to adapt commercial motion tracking controllers and visual feedback into engaging rehabilitative learning tools. This study will focus on a basic science aspect of human bimanual movements that can be incorporated into future applications of the full FEATHERS project devices. We believe that together these approaches will yield interventions that significantly improve functional ability and lead to improved quality of life.

DETAILED DESCRIPTION:
(Main Phase Only - Data Collected with Clinical Population)

The FEATHERS project at the RREACH Lab at The University of British Columbia focuses on developing and evaluating novel physical exercise technologies for kids with motor disabilities. The study team would like to study how immersive virtual reality (VR) technology can be used to benefit upper limb rehabilitation for persons with hemiplegia. The purpose of the experiment is to see how the use of error augmentation (i.e. adding visual or game element feedback to accentuate deviation from the desired exercise motion) might encourage persons with hemiplegia to engage their affected side more effectively by comparing the symmetry between the stronger and weaker limbs. It is also hypothesized that the immersive environment of VR and the ability to provide 1:1 direct visual feedback will increase active engagement to rehabilitative exercises in these populations. The study will address the question of whether error augmentation aids in the rehabilitation of the affected upper limb movement quality in hemiparesis when practicing bilateral reaching tasks. Specifically, can visual amplification of paretic asymmetry in an immersive VR environment improve movement quality in the affected side?

Adolescents and young adults with hemiplegia (i.e. due to ABI, CP, etc.) and their adjoining therapists will be recruited for from the community. We will conduct testing in a single-session setup at the participant chosen location with an easily transportable system including a standard 2-3 sensor Oculus system hardware setup and software developed by the research team. Sessions conducted outside the research lab rooms will require a minimum of a 2m x 1.5m space for calibration. The participants will test all augmentation factors in a randomized order and the sessions are expected to take between 90-120 minutes. A short post-session usability survey will be administered and sample population demographic data will be recorded including age, gender, and handedness. Manual Ability Classification System (MACS) and Bimanual Fine Motor Function (BFMF) scores will be recorded or assessed to classify the upper limb motor ability of the sample set.

ELIGIBILITY:
Inclusion for adolescents and young adults (ages 13-21 years) :

i. Hemiplegia as a result of a neurological impairment (CP, ABI, paediatric stroke, etc.)

ii. Use both eyes and visually interact using a stereoscopic device that allows a minimum interpupillary distance of 58mm

iii. Comfortably support regular head motion while wearing a 470g head-mounted display

iv. Ability to lift arms against gravity at least some distance away from their body (some shoulder and elbow flexion and extension) as reported by participant, consenting guardian, or adjoining therapist

v. Ability to stand or sit independently for 15 minutes at a time in a chair without arm supports for a total of up to 120 minutes

vi. Ability to follow instructions and verbally communicate in basic English (as determined by referring therapist)

Exclusion Criteria:

i. Upper limb orthopedic surgery in the past six months

ii. Known susceptibility to cybersickness

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Change in Error in Forward Reaching Symmetry | Recorded per reach, throughout the session (about 2 hours)
  Compared between each condition (in cm, % change from baseline)

SECONDARY OUTCOMES:
Distance traveled of each arm from head | Recorded per reach, throughout the session (about 2 hours)
  Change in position in cm of the participant hands from the start to end of the reach trial
Time to complete task | Recorded per reach, throughout the session (about 2 hours)
  Time in seconds from the start to the end of the reach trial
Movement Smoothness | Recorded per arm, per reach, throughout the session (about 2 hours)
  Deviation from linear path in the lateral direction and number of peaks in forward velocity profile
Change in Error in Forward Reaching Symmetry Over Time | Recorded per reach, throughout the session (about 2 hours)
  Change in error throughout each set during the learning conditions
Compensation Techniques Causing Joint Asymmetry | Recorded throughout the session (about 2 hours)
  Maximum difference in cm in contralateral joint position in the upper body (shoulder y, z)
Trunk Compensation | Recorded throughout the session (about 2 hours)
  Change in forward position in cm of the participant head and trunk (mid-shoulder point) during reaching movement

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik FM Van der Loos, PhD, P.Eng, Principal Investigator — The University of British Columbia
Locations (2):
- Canada (2):
  - Physiotherapy, BC Children's Hospital, Vancouver, British Columbia
  - RREACH Lab, The University of British Columbia, Vancouver, British Columbia

REFERENCES:
- [Derived] Shum LC, Valdes BA, Hodges NJ, Van der Loos HFM. Error Augmentation in Immersive Virtual Reality for Bimanual Upper-Limb Rehabilitation in Individuals With and Without Hemiplegic Cerebral Palsy. IEEE Trans Neural Syst Rehabil Eng. 2020 Feb;28(2):541-549. doi: 10.1109/TNSRE.2019.2959621. Epub 2019 Dec 13. PMID 31841417